CLINICAL TRIAL: NCT04211597
Title: EGF-loaded Chitosan to Facilitate Epithelial Healing And Prevent Scar Formation of Cesarean Wound
Brief Title: EGF-loaded Chitosan to Facilitate Healing and Prevent Scar Formation of Cesarean Wound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, TING-CHANG CHANG, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201601310A3
Record Dates: First submitted 2019-12-20; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Cesarean Wound; Scar; Previous Cesarean Section, Complicating Pregnancy or Childbirth, Affecting Fetus or Newborn
MeSH Terms: conditions — Cicatrix; Pregnancy Complications | interventions — Silicone Gels

STUDY DESIGN:
Intervention Model Description: Upon enrollment, full medical history of the participants was obtained, including history of hypertrophic scar or keloid. Scars from previous injuries or surgical incisions were evaluated and recorded. Each patient was randomized to one of the three treatment arms: Group 1 (receiving no scar treatment), Group 2 (silicone gel only), and Group 3 (silicone gel plus Me-EGF).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the distinctive nature between types of scar treatments (spray vs gel, or no treatment at all), care provider and patients will not be blind to the group assignment. However, outcomes assessors are trained nurse practitioners and research associates, who do not have access to participants' group assignment records.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Control (Sham Comparator): Participants receive no scar prevention and treatment for Cesarean wounds.
  Interventions: Other: Control
- Group 2: Silicone gel (Active Comparator): Each participant in Group 2 brought home two tubes of silicone gel when they returned for their follow-up visits on day 14. They were instructed to start applying silicone gel evenly to the wound twice a day for two months.
  Interventions: Other: Silicone gel
- Group 3: Silicone gel plus Me-EGF (Experimental): 1. The day of Cesarean delivery was recorded as Day 0. For participants in Group 3, on day 0 prior to final dermal closure, 4ml of Me-EGF (containing 40mcg microencapsulated polysaccharide and rhEGF) was sprayed evenly along the incision site, subsequently covered with antibiotic ointment and sterile gauze. Another 0.5 ml (5 mcg of Me-EGF) was sprayed during dressing change on day 1 and day 5 respectively. At each dressing change, the sutured wound was cleaned by sterile normal saline, followed by Me-EGF sprays, and waited for two minutes to allow for absorption, then covered with dry sterile gauze.
  2. Each participant in Group 3 brought home two tubes of silicone gel when they returned for their follow-up visits on day 14. They were instructed to start applying silicone gel evenly to the wound twice a day for two months.
  Interventions: Other: Silicone gel; Other: microencapsulated polysaccharide and oligopeptide-1(Me-EGF) 40 mcg & 5 mcg

INTERVENTIONS:
Other: Control — No scar prevention or treatment.
  Arms: Group 1: Control
Other: Silicone gel — Dermatix® (Dermatix® Ultra, Menarini Asia-Pacific, Taiwan FDA approved)
  Arms: Group 2: Silicone gel; Group 3: Silicone gel plus Me-EGF
Other: microencapsulated polysaccharide and oligopeptide-1(Me-EGF) 40 mcg & 5 mcg — 4ml (40 mcg) of Me-EGF spray will be given by the operating physician prior to wound closure, followed by daily application of 5 mcg until day +5 after delivery. Starting from day +14, participants will receive FDA approved Silicone gel to be applied to the Cesarean wound twice a day for two months. Participants also receive routine post-partum care as usual.
  Arms: Group 3: Silicone gel plus Me-EGF

SUMMARY:
Cesarean section (CS) is a major surgical intervention that affects women at childbearing age. Scarring from CS potentially causes discomfort and psychological distress. Emerging evidence indicates that epidermal growth factor (EGF) plays crucial roles in wound healing with the potential of minimizing scar formation. This study aims to investigate the effect of microencapsulated recombinant human EGF (Me-EGF) in scar prevention. Silicone gel was incorporated as part of the routine scar treatment.

Healthy women scheduled for cesarean delivery will be enrolled and randomized to three groups: (1) no scar treatment, (2) silicone gel only, or (3) silicone gel plus Me-EGF. Vancouver Scar Scale (VSS) will be used for scar assessment at the 6th month and 9th month after CS.

DETAILED DESCRIPTION:
Objective:

Cesarean section (CS) is a major surgical intervention that affects women at childbearing age. Scarring from CS is expected but certainly not desirable, potentially causes discomfort and psychological distress. Emerging evidence indicates that epidermal growth factor (EGF) plays crucial roles in wound healing with the potential of minimizing scar formation. This study aims to investigate the effect of microencapsulated recombinant human EGF (Me-EGF) in scar prevention. Silicone gel was incorporated as part of the routine scar treatment.

Materials:

The investigational dressing in this study: the microencapsulated polysaccharide and oligopeptide-1 is provided by Good-Care Biotech, Ltd. (brand NewEpi®: 10 mcg Me-EGF/ml, Taipei, Taiwan). The investigational dressing NewEpi® was formulated in spray solution with a proprietary drug delivery system in which rhEGF was encapsulated in chitosan as nanoparticles.

Silicone-based scar therapy has shown the beneficial effects of improving the appearance of scars. Dermatix® (Dermatix® Ultra, Menarini Asia-Pacific, Taiwan) is a Taiwan-FDA approved topical silicone gel and commercially available. It is transparent, odorless and quick drying. Concerning the applicability over lower abdomen area, silicone gel (Dermatix®) was selected to be part of the routine care in this study.

Study Procedures:

Healthy women scheduled for cesarean delivery were enrolled and randomized to three groups: (1) no scar treatment, (2) silicone gel only, or (3) silicone gel plus Me-EGF. Vancouver Scar Scale (VSS: vascularity, pigmentation, elasticity, and height) was used for scar assessment at the 6th month and 9th month after CS.

Eligibility was determined at the screening visit. Details of the study regarding eligibility, purpose, study procedure, scope of care and potential risks were explained. Upon enrollment, full medical history of the participants was obtained, including history of hypertrophic scar or keloid. Scars from previous injuries or surgical incisions were evaluated and recorded. Each patient was randomized to one of the three treatment arms: Group 1 (receiving no scar treatment), Group 2 (silicone gel only), and Group 3 (silicone gel plus Me-EGF). Enrolled participants underwent Cesarean delivery performed by one of the four obstetricians at the Department of Obstetrics and Gynecology of CGMH, as part of their prenatal care. Other than routine surgical wound care, participants in Group 1 did not receive any treatment pertaining to scar prevention.

The day of Cesarean delivery was recorded as Day 0. For participants in Group 3, on day 0 prior to final dermal closure, 4ml of Me-EGF (containing 40mcg microencapsulated polysaccharide and rhEGF) was sprayed evenly along the incision site, subsequently covered with antibiotic ointment and sterile gauze. Another 0.5 ml (5 mcg of Me-EGF) was sprayed during dressing change on day 1 and day 5 respectively. At each dressing change, the sutured wound was cleaned by sterile normal saline, followed by Me-EGF sprays, and waited for two minutes to allow for absorption, then covered with dry sterile gauze. Each participant in Group 2 and Group3 brought home two tubes of silicone gel when they returned for their follow-up visits on day 14. They were instructed to start applying silicone gel evenly to the wound twice a day for two months.

Study Participants:

This study is approved by the Institutional Review Board at Chang-Gung Memorial Hospital (CGMH, Linkou, Taiwan). All practitioners and research staffs are in compliance with Good Clinical Practice guidelines. A total of 60 females scheduled for cesarean birth will be recruited by their primary obstetricians at the Department of Obstetrics and Gynecology of CGMH. Prior to their enrollment, the study procedures will be explained to obtain written informed consents. The inclusion criteria are: (1) Age of 18 or older; (2) planned for cesarean delivery with Pfannenstiel-incision, which is one common method of performing Caesarian sections today; (3) had not received any treatment for scars at least one month before enrollment; and (4) capable of understanding study protocol in order to sign the informed consent voluntarily.

Patients will be excluded if: (1) currently taking any medication that might affect outcome evaluation of this study, including but not limited to: systemic corticosteroids or immunosuppressants; (2) currently undergoing any treatments involving lower abdomen, or planning to have such treatments; (3) having active infection involving abdomen at the time of recruitment; (4) concomitant severe or poorly-controlled illness (e.g., cardiovascular, renal, hepatic, pulmonary or gastrointestinal disease, malignancy or history of HIV infection); (5) with any abdominal tumor; (6) undergoing urgent cesarean delivery without proper pre-op standard procedure, or (7) having known allergy to any of the ingredients in any of the products used in this study.

Clinical Evaluation and Outcome Measures:

There were a total of four time points at which data were collected and photos taken using the same digital camera with fixed settings: day 0 (completion of suture on Cesarean incision), day 1, day 5 before discharge from the hospital, and at follow-up visits in month 3, month 6, and month 9. After enrollment and before day 0, baseline photos of old Cesarean scars were taken from participants who had prior Cesarean childbirth, in addition to photos of other scars from those who had reported history of hypertrophic scar or keloid. Scars were assessed using Vancouver Scar Scale. The VSS consists of 4 parameters: vascularity (0-3), pigmentation (0-3), elasticity (0-5), and height (0-3). Prior to the study commencement, all personnel involved had received mandatory training on scar assessment and VSS scoring. At month 3, 6, and 9, a nurse practitioner took photos and evaluated the incision scar on each patient with VSS. Photos of each healing wound were taken with a ruler placed adjacent to the scar to measure the height raised above skin level. Subsequently all scores were validated twice by different research staffs by using the photos on record. No significant discrepancies were found. At each follow-up visit, the primary obstetrician also assessed each patient for any side effect or adverse event.

Statistical Analysis:

Clinical data and all scar measurements were recorded on case report forms and entered in Microsoft Excel database, later validated by different research staffs as the final scores. Data were analyzed using jamovi statistical software (Version 0.9). Means and standard deviations were presented for interval variables of baseline characteristics. Categorical data at baseline were presented in frequency and analyzed with Chi-Square tests. Nonparametric Kruskal-Wallis tests were performed on VSS scores for between group comparisons. A p-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older
* Planned for cesarean delivery with Pfannenstiel-incision
* Had not received any treatment for scars at least one month before enrollment
* Capable of understanding study protocol in order to sign the informed consent voluntarily

Exclusion Criteria:

* Currently taking any medication that might affect outcome evaluation of this study, including but not limited to: systemic corticosteroids or immunosuppressants
* Currently undergoing any treatments involving lower abdomen, or planning to have such treatments
* Having active infection involving abdomen at the time of recruitment
* Concomitant severe or poorly-controlled illness (e.g., cardiovascular, renal, hepatic, pulmonary or gastrointestinal disease, malignancy or history of HIV infection)
* With any abdominal tumor
* Undergoing urgent cesarean delivery without proper pre-op standard procedure
* Having known allergy to any of the ingredients in any of the products used in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Vascularity | Evaluation of Vascularity is done at: month 3+ follow-up visit.
  Vascularity is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Pink; 2: Red; 3: Purple
Pigmentation | Evaluation of Pigmentation is done at: month 3+ follow-up visit.
  Vascularity is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Hypo-pigmentation; 2: Mixed-pigmentation; 3: Hyper-pigmentation
Pliability | Evaluation of Pliability is done at: month 3+ follow-up visit.
  Pliability is one the the four subscales in Vancouver Scar Scale (VSS). Score range: 0-5. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Supple; 2: Yielding; 3: Firm; 4: Banding; 5: Contracture
Height | Evaluation of Height is done at: month 3+ follow-up visit.
  Height of the scar is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: flat; 1: 0-2mm; 2: 2-5mm; 3: > 5mm
Vascularity | Evaluation of Vascularity is done at: month 6+ follow-up visit.
  Vascularity is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Pink; 2: Red; 3: Purple
Pigmentation | Evaluation of Pigmentation is done at: month 6+ follow-up visit.
  Vascularity is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Hypo-pigmentation; 2: Mixed-pigmentation; 3: Hyper-pigmentation
Pliability | Evaluation of Pliability is done at: month 6+ follow-up visit.
  Pliability is one the the four subscales in Vancouver Scar Scale (VSS). Score range: 0-5. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Supple; 2: Yielding; 3: Firm; 4: Banding; 5: Contracture
Height | Evaluation of Height is done at: month 6+ follow-up visit.
  Height of the scar is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: flat; 1: 0-2mm; 2: 2-5mm; 3: > 5mm
Vascularity | Evaluation of Vascularity is done at: month 9+ follow-up visit.
  Vascularity is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Pink; 2: Red; 3: Purple
Pigmentation | Evaluation of Pigmentation is done at: month 9+ follow-up visit.
  Vascularity is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Hypo-pigmentation; 2: Mixed-pigmentation; 3: Hyper-pigmentation
Pliability | Evaluation of Pliability is done at: month 9+ follow-up visit.
  Pliability is one the the four subscales in Vancouver Scar Scale (VSS). Score range: 0-5. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: Normal; 1: Supple; 2: Yielding; 3: Firm; 4: Banding; 5: Contracture
Height | Evaluation of Height is done at: month 9+ follow-up visit.
  Height of the scar is one of the four subscales in Vancouver Scar Scale (VSS). Score range: 0-3. It is a Likert-type scale of which score 0 indicates normal or none, and a higher score indicates the severity of the specific condition. Assessed at 3 time points: Month 3+, Month 6+ and Month 9+ postpartum visits. A trained nurse practitioner evaluates participant's Cesarean wound scar and assigns a score when the participant returns to the follow-up appointment.
  0: flat; 1: 0-2mm; 2: 2-5mm; 3: > 5mm

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Kirsner RS, Eaglstein WH. The wound healing process. Dermatol Clin. 1993 Oct;11(4):629-40. PMID 8222347
- [Background] O'Kane S, Ferguson MW. Transforming growth factor beta s and wound healing. Int J Biochem Cell Biol. 1997 Jan;29(1):63-78. doi: 10.1016/s1357-2725(96)00120-3. PMID 9076942
- [Background] Shah M, Foreman DM, Ferguson MW. Neutralisation of TGF-beta 1 and TGF-beta 2 or exogenous addition of TGF-beta 3 to cutaneous rat wounds reduces scarring. J Cell Sci. 1995 Mar;108 ( Pt 3):985-1002. doi: 10.1242/jcs.108.3.985. PMID 7542672
- [Background] Peled ZM, Rhee SJ, Hsu M, Chang J, Krummel TM, Longaker MT. The ontogeny of scarless healing II: EGF and PDGF-B gene expression in fetal rat skin and fibroblasts as a function of gestational age. Ann Plast Surg. 2001 Oct;47(4):417-24. doi: 10.1097/00000637-200110000-00010. PMID 11601578
- [Background] Satici A, Guzey M, Dogan Z, Kilic A. Relationship between Tear TNF-alpha, TGF-beta1, and EGF levels and severity of conjunctival cicatrization in patients with inactive trachoma. Ophthalmic Res. 2003 Nov-Dec;35(6):301-5. doi: 10.1159/000074067. PMID 14688418
- [Background] Kim YS, Lew DH, Tark KC, Rah DK, Hong JP. Effect of recombinant human epidermal growth factor against cutaneous scar formation in murine full-thickness wound healing. J Korean Med Sci. 2010 Apr;25(4):589-96. doi: 10.3346/jkms.2010.25.4.589. Epub 2010 Mar 19. PMID 20358003
- [Background] Ferguson MW, Duncan J, Bond J, Bush J, Durani P, So K, Taylor L, Chantrey J, Mason T, James G, Laverty H, Occleston NL, Sattar A, Ludlow A, O'Kane S. Prophylactic administration of avotermin for improvement of skin scarring: three double-blind, placebo-controlled, phase I/II studies. Lancet. 2009 Apr 11;373(9671):1264-74. doi: 10.1016/S0140-6736(09)60322-6. PMID 19362676
- [Background] Repertinger SK, Campagnaro E, Fuhrman J, El-Abaseri T, Yuspa SH, Hansen LA. EGFR enhances early healing after cutaneous incisional wounding. J Invest Dermatol. 2004 Nov;123(5):982-9. doi: 10.1111/j.0022-202X.2004.23478.x. PMID 15482488
- [Background] Brown GL, Curtsinger LJ, White M, Mitchell RO, Pietsch J, Nordquist R, von Fraunhofer A, Schultz GS. Acceleration of tensile strength of incisions treated with EGF and TGF-beta. Ann Surg. 1988 Dec;208(6):788-94. doi: 10.1097/00000658-198812000-00019. PMID 3264140
- [Background] Shin JU, Kang SW, Jeong JJ, Nam KH, Chung WY, Lee JH. Effect of recombinant human epidermal growth factor on cutaneous scar quality in thyroidectomy patients. J Dermatolog Treat. 2015 Apr;26(2):159-64. doi: 10.3109/09546634.2014.906034. Epub 2014 Apr 8. PMID 24708156
- [Background] Lee DW, Lim C, Israelachvili JN, Hwang DS. Strong adhesion and cohesion of chitosan in aqueous solutions. Langmuir. 2013 Nov 19;29(46):14222-9. doi: 10.1021/la403124u. Epub 2013 Nov 6. PMID 24138057
- [Background] Lim C, Lee DW, Israelachvili JN, Jho Y, Hwang DS. Contact time- and pH-dependent adhesion and cohesion of low molecular weight chitosan coated surfaces. Carbohydr Polym. 2015 Mar 6;117:887-894. doi: 10.1016/j.carbpol.2014.10.033. Epub 2014 Nov 5. PMID 25498713
- [Background] Mao S, Sun W, Kissel T. Chitosan-based formulations for delivery of DNA and siRNA. Adv Drug Deliv Rev. 2010 Jan 31;62(1):12-27. doi: 10.1016/j.addr.2009.08.004. Epub 2009 Sep 29. PMID 19796660
- [Background] Chan KY, Lau CL, Adeeb SM, Somasundaram S, Nasir-Zahari M. A randomized, placebo-controlled, double-blind, prospective clinical trial of silicone gel in prevention of hypertrophic scar development in median sternotomy wound. Plast Reconstr Surg. 2005 Sep 15;116(4):1013-20; discussion 1021-2. doi: 10.1097/01.prs.0000178397.05852.ce. PMID 16163087
- [Background] Chernoff WG, Cramer H, Su-Huang S. The efficacy of topical silicone gel elastomers in the treatment of hypertrophic scars, keloid scars, and post-laser exfoliation erythema. Aesthetic Plast Surg. 2007 Sep-Oct;31(5):495-500. doi: 10.1007/s00266-006-0218-1. PMID 17700980
- [Background] Signorini M, Clementoni MT. Clinical evaluation of a new self-drying silicone gel in the treatment of scars: a preliminary report. Aesthetic Plast Surg. 2007 Mar-Apr;31(2):183-7. doi: 10.1007/s00266-005-0122-0. PMID 17171514
- [Background] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427
- [Background] Tyack Z, Simons M, Spinks A, Wasiak J. A systematic review of the quality of burn scar rating scales for clinical and research use. Burns. 2012 Feb;38(1):6-18. doi: 10.1016/j.burns.2011.09.021. Epub 2011 Nov 1. PMID 22047828
- [Result] Reinke JM, Sorg H. Wound repair and regeneration. Eur Surg Res. 2012;49(1):35-43. doi: 10.1159/000339613. Epub 2012 Jul 11. PMID 22797712
- [Result] Baum CL, Arpey CJ. Normal cutaneous wound healing: clinical correlation with cellular and molecular events. Dermatol Surg. 2005 Jun;31(6):674-86; discussion 686. doi: 10.1111/j.1524-4725.2005.31612. PMID 15996419
- [Result] Mustoe TA, Cooter RD, Gold MH, Hobbs FD, Ramelet AA, Shakespeare PG, Stella M, Teot L, Wood FM, Ziegler UE; International Advisory Panel on Scar Management. International clinical recommendations on scar management. Plast Reconstr Surg. 2002 Aug;110(2):560-71. doi: 10.1097/00006534-200208000-00031. PMID 12142678
- [Result] McCarty M. An evaluation of evidence regarding application of silicone gel sheeting for the management of hypertrophic scars and keloids. J Clin Aesthet Dermatol. 2010 Nov;3(11):39-43. No abstract available. PMID 21103316
- [Result] Mustoe TA. Evolution of silicone therapy and mechanism of action in scar management. Aesthetic Plast Surg. 2008 Jan;32(1):82-92. doi: 10.1007/s00266-007-9030-9. Epub 2007 Oct 30. PMID 17968615
- [Result] Borgognoni L. Biological effects of silicone gel sheeting. Wound Repair Regen. 2002 Mar-Apr;10(2):118-21. doi: 10.1046/j.1524-475x.2002.00205.x. No abstract available. PMID 12028528
- [Result] Stavrou D. Neovascularisation in wound healing. J Wound Care. 2008 Jul;17(7):298-300, 302. doi: 10.12968/jowc.2008.17.7.30521. PMID 18705231
- [Result] Perry DM, McGrouther DA, Bayat A. Current tools for noninvasive objective assessment of skin scars. Plast Reconstr Surg. 2010 Sep;126(3):912-923. doi: 10.1097/PRS.0b013e3181e6046b. PMID 20811225
- [Result] Idriss N, Maibach HI. Scar assessment scales: a dermatologic overview. Skin Res Technol. 2009 Feb;15(1):1-5. doi: 10.1111/j.1600-0846.2008.00327.x. PMID 19152571
- [Result] Micallef L, Vedrenne N, Billet F, Coulomb B, Darby IA, Desmouliere A. The myofibroblast, multiple origins for major roles in normal and pathological tissue repair. Fibrogenesis Tissue Repair. 2012 Jun 6;5(Suppl 1):S5. doi: 10.1186/1755-1536-5-S1-S5. eCollection 2012. PMID 23259712
- [Result] Kelly AP. Medical and surgical therapies for keloids. Dermatol Ther. 2004;17(2):212-8. doi: 10.1111/j.1396-0296.2004.04022.x. PMID 15113289
- [Result] Anzarut A, Olson J, Singh P, Rowe BH, Tredget EE. The effectiveness of pressure garment therapy for the prevention of abnormal scarring after burn injury: a meta-analysis. J Plast Reconstr Aesthet Surg. 2009 Jan;62(1):77-84. doi: 10.1016/j.bjps.2007.10.052. Epub 2008 Jan 14. PMID 18249046
- [Result] Xue M, Jackson CJ. Extracellular Matrix Reorganization During Wound Healing and Its Impact on Abnormal Scarring. Adv Wound Care (New Rochelle). 2015 Mar 1;4(3):119-136. doi: 10.1089/wound.2013.0485. PMID 25785236
- [Result] Bond JS, Duncan JAL, Sattar A, Boanas A, Mason T, O'Kane S, Ferguson MWJ. Maturation of the human scar: an observational study. Plast Reconstr Surg. 2008 May;121(5):1650-1658. doi: 10.1097/PRS.0b013e31816a9f6f. PMID 18453989
- [Result] Chang CW, Ries WR. Nonoperative techniques for scar management and revision. Facial Plast Surg. 2001 Nov;17(4):283-8. doi: 10.1055/s-2001-18826. PMID 11735062
- [Result] Berlanga-Acosta J, Gavilondo-Cowley J, Lopez-Saura P, Gonzalez-Lopez T, Castro-Santana MD, Lopez-Mola E, Guillen-Nieto G, Herrera-Martinez L. Epidermal growth factor in clinical practice - a review of its biological actions, clinical indications and safety implications. Int Wound J. 2009 Oct;6(5):331-46. doi: 10.1111/j.1742-481X.2009.00622.x. PMID 19912390